CLINICAL TRIAL: NCT01023568
Title: Comparison of Direct Laryngoscopy, Truview EVO2 and Glidescope in Pediatric Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped for futility at the first interim analysis
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 09-902
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Intubation
Keywords: intubation; pediatric; videolaryngoscope devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Macintosh blade (Active Comparator): Intubation with Macintosh blade laryngoscope
  Interventions: Device: Macintosh blade
- Glidescope (Active Comparator): Intubation with Glidescope laryngoscope
  Interventions: Device: Glidescope
- Truview PCD (Active Comparator): Intubation with the Truview PCD laryngoscope
  Interventions: Device: Truview PCD

INTERVENTIONS:
Device: Macintosh blade — Intubation with Macintosh blade laryngoscope
  Arms: Macintosh blade
Device: Glidescope — Intubation with Glidescope laryngoscope.
  Arms: Glidescope
Device: Truview PCD — Intubation with Truview PCD laryngoscope.
  Arms: Truview PCD

SUMMARY:
The purpose of this study is to compare the effectiveness of two novel videolaryngoscope systems, the Glidescope and the Truview PCD against standard direct laryngoscopy (DL) in pediatric patients. The investigators primary hypothesis is that the use of videolaryngoscope devices, Glidescope and Truview provide better laryngeal views in pediatric patients as measured by Cormack and ehane (C&L) (1 to 4, 4 the worst), without increasing the time taken to intubate (TTI), compared with direct laryngoscopy (DL).

The investigators secondary hypotheses are that the use of Glidescope and Truview PCD provoke less hemodynamic response and fewer episodes of de-saturation in pediatric patients.

DETAILED DESCRIPTION:
Advances in airway management have led to development on videolaryngoscopy devices including the Glidescope® (Verathon Inc, Bothwell, USA), the AWD® (Pentax Corporation, Tokio, Japan) and most recently the Truview PCD (Truphatek International Ltd, Netanya, Israel). The use of videolaryngoscopy devices in adults have demonstrated some advantages including, minimal trauma on the airway and better view of the glottis.

The Glidescope is designed with a 60º angle and a camera on the inferior aspect just at the inflection point. The view is obtained anteriorly and the camera is located remote from the glottis providing a good visual field. The video image is displayed on a Liquid Crystal Display (LCD), with electronic recording available. Despite a good experience using Glidescope in adults, few studies have been published in pediatric patients. Kim et al. in a randomized study comparing the use of Glidescope with direct laryngoscopy in children, demonstrated better or equal laryngoscopic view with longer time for intubation using the Glidescope.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* elective general surgical procedures
* from 0-10 years-old

Exclusion Criteria:

* increase intracranial pressure
* history of severe gastrointestinal reflux
* sore throat
* upper respiratory airway infection
* known or suspected difficult airway or coagulopathy

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2009-12; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Niezgoda, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Macintosh Blade | Glidescope | Truview PCD
Started | 45 | 44 | 45
Completed | 45 | 44 | 45
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Macintosh Blade | Glidescope | Truview PCD | Total
Number analyzed (Participants) | 45 | 44 | 45 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.0 (2.8) | 4.6 (2.7) | 5.2 (2.8) | 4.6 (2.8)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 11 | 14 | 41
  Male | 29 | 33 | 31 | 93
Body mass index [Median (Inter-Quartile Range); unit: kg/m2] | 17 [15 to 19] | 16 [15 to 18] | 16 [16 to 18] | 16.5 [15.4 to 18.8]
ASA physical status [Number; unit: participants]
  I: A normal healthy patient | 19 | 20 | 19 | 58
  II: A patient with mild systemic disease | 24 | 23 | 25 | 72
  III: A patient with severe systemic disease | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Successfully Intubate Patient.
Time Frame: from start of intubation to successfully intubated up to 5 minutes
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Macintosh Blade | Glidescope | Truview PCD
Number analyzed (Participants) | 45 | 44 | 45
seconds | 23 [21 to 28] | 39 [31 to 59] | 44 [28 to 62]
Statistical Analysis 1: Comparison: Macintosh Blade vs Glidescope; Test type: Non-Inferiority or Equivalence — The GlideScope and Truview PCD video laryngoscopes were individually assessed for non-inferiority on time to intubation vs direct laryngoscopy at the 0.025 significance level using an a priori specified non-inferiority delta of seven seconds (about 40% of the expected standard deviation of 18 sec and not thought to be clinically important); p > 0.99, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 14, 95% CI 2-sided [7 to 26] — Glidescope - direct laryngoscopy
Statistical Analysis 2: Comparison: Macintosh Blade vs Truview PCD; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p > 0.99, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 17, 95% CI 2-sided [6 to 28] — Truview PCD - direct laryngoscopy

2. Secondary Outcome: Mean Hemodynamic Response: Mean Arterial Blood Pressure
Time Frame: measured at 1 minute interval at induction time and from intubation for 10 minutes
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Macintosh Blade | Glidescope | Truview PCD
Number analyzed (Participants) | 45 | 44 | 45
mmHg | 62 (12) | 63 (9) | 66 (12)
Statistical Analysis 1: Comparison: Macintosh Blade vs Glidescope vs Truview PCD; Test type: Superiority or Other; p = 0.28, ANOVA

3. Secondary Outcome: Cormack-Lehane Grade
Time Frame: immediately after intubation
Measure: Number; unit: participants
Arm/Group | Macintosh Blade | Glidescope | Truview PCD
Number analyzed (Participants) | 45 | 44 | 45
participants
  1: Full view of glottis | 34 | 6 | 37
  2: Partial view of glottis | 6 | 13 | 7
  3: Only epiglottis seen, none of glottis seen | 5 | 23 | 1
  4: Neither glottis nor epiglottis seen | 0 | 2 | 0
Statistical Analysis 1: Comparison: Macintosh Blade vs Glidescope; The Cormack-Lehane grade with a grade 1 (best grade) to 4 (worst grade) was analyzed as an ordinal outcome; Test type: Superiority or Other; p > 0.99, Wilcoxon (Mann-Whitney); 1-tailed Wilcoxon sum-rank test; Median Difference (Final Values) = 1, 95% CI 2-sided [1 to 2] — The median difference was Hodges-Lehmann estimation and the confidence intervals were exact confidence limits. The SAS "NPAR1WAY" procedure was used for test and estimation
Statistical Analysis 2: Comparison: Macintosh Blade vs Truview PCD; The Cormack-Lehane grade with a grade 1 (best grade) to 4 (worst grade) was analyzed as an ordinal outcome; Test type: Superiority or Other; p = 0.18, Wilcoxon (Mann-Whitney); 1-tailed Wilcoxon sum-rank test; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Mean Hemodynamic Response: Heart Rate
Time Frame: measured at 1 minute interval at induction time and from intubation for 10 minutes.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Macintosh Blade | Glidescope | Truview PCD
Number analyzed (Participants) | 45 | 44 | 45
beats/min | 126 (21) | 127 (15) | 128 (18)
Statistical Analysis 1: Comparison: Macintosh Blade vs Glidescope vs Truview PCD; Test type: Superiority or Other; p = 0.26, ANOVA

5. Secondary Outcome: Number of Participants Who Experienced Desaturation
Description: Desaturation was defined as SpO2 less than 90% at induction time or any time from intubation to 10 minutes after
Time Frame: measured at 1 minute interval at induction time and from intubation for 10 minutes.
Measure: Number; unit: participants
Arm/Group | Macintosh Blade | Glidescope | Truview PCD
Number analyzed (Participants) | 45 | 44 | 45
participants | 1 | 0 | 1
Statistical Analysis 1: Comparison: Macintosh Blade vs Glidescope vs Truview PCD; Test type: Superiority or Other; p > 0.99, Chi-squared

ADVERSE EVENTS:
Arm/Group | Macintosh Blade | Glidescope | Truview PCD
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/44 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No